CLINICAL TRIAL: NCT02157831
Title: Redosing With CP-870,893 in Patients With Clinical Benefit After a Single Infusion of CP-870,893 From A Phase I, Open-Label, Dose-Escalation Study of CP-870,893 in Patients With Solid Tumors
Brief Title: Redosing With CP-870, 893 in Patients With Clinical Benefit After a Single Infusion From A Phase I, Open-Label, Dose-Escalation Study of CP-870,893 in Patients With Solid Tumors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: UPCC 10904
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Solid Tumors
Keywords: Subjects with Clinical Benefit After a Single Infusion of CP - 870, 893
MeSH Terms: interventions — selicrelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Subjects from UPCC 10903 (Experimental)
  Interventions: Biological: CP-870,893

INTERVENTIONS:
Biological: CP-870,893

SUMMARY:
Patients who had clinical benefit following a single infusion of CP-870, 893 on Protocol UPCC 10903 will receive a single repeated infusion of CP-870,893 at the same dose given on UPCC 10903 intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Clinical benefit, including stable disease, partial response, or complete response, without a dose-limiting toxicity after a single infusion of CP-870,893; however, patients who experienced transient, not serious, and fully reversible grade 1-3 increases in ALT or AST after one dose of CP-870,893 may, if otherwise eligible, receive a second dose on this protocol.
* Age at least 18 years old;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1;
* Adequate bone marrow function documented within 2 weeks prior to treatment, defined as:
* White blood cell (WBC) count >3000 cells/μL without growth factor support;
* Absolute neutrophil count (ANC) ≥1500/μL without growth factor support;
* Platelets >100,000/μL without growth factor support; and
* Hemoglobin ≥10 g/dL.
* Adequate renal and hepatic function documented within 2 weeks prior to treatment, defined as:
* Total bilirubin <1.5 times the upper limit of normal (ULN);
* Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) <2.5 × ULN;
* Creatinine clearance (CLcr, measured or calculated) >80 mL/min; and
* Life expectancy of at least 12 weeks;
* Signed written informed consent.

Exclusion Criteria

* Concurrent treatment with any anticancer agent;
* History of autoimmune disorder, including pemphigus vulgaris, systemic mastocytosis, systemic lupus erythamatosus, dermatomyositis/polymyositis, rheumatoid arthritis, systemic sclerosis, Sjörgen's syndrome, vasculitis/arteritis, Behcet's syndrome, inflammatory bowel disease, autoimmune thyroiditis, multiple sclerosis, or other chronic inflammatory disease;
* Treatment with any other cancer therapy from the time of the first dose of CP-870,893, except as noted in Section 4.4; 1 Cancer Therapy Evaluation Program, Common Terminology Criteria for Adverse Events, Version 3.0, DCTD, NCI, NIH, DHHS. 31 Mar 2003 (http://ctep.cancer.gov).
* History of congestive heart failure, stroke, or myocardial infarction;
* Hereditary or acquired coagulopathies (e.g. hemophilia, von Willebrand's disease, cancer-associated DIC);
* Brain metastases.
* Patient having reproductive potential who is not using an effective method of birth control or who is pregnant or breastfeeding or has a positive (urine or serum) pregnancy test at baseline;
* Known sensitivity to immunomodulating agents or monoclonal antibodies;
* Alcohol abuse or illicit drug use within 12 months of enrollment;
* History of serum creatinine ≥2 mg/dL for any duration and for any reason;
* Urine dipstick 1+ or more positive for blood (other than menstruating females) or 2+ or more positive for protein;
* Positive HAHA antibody titer in response to treatment with first dose of CP-870,893 (as determined by Pfizer)
* Clinically significant presence of granular or cellular casts in centrifuged urine sediment;
* Renal carcinoma or renal metastases;
* Partial or complete nephrectomy;
* History of dialysis (peritoneal or hemodialysis);
* Prior treatment with Amphotericin B or cisplatin;
* History of insulin-dependent diabetes for greater than 5 years;
* Concomitant treatment with systemic corticosteroids or treatment with systemic corticosteroids within 4 weeks of baseline;
* Concomitant treatment with anticoagulants, such as coumadin or heparin, except to maintain patency of in-dwelling catheters;
* Prior allergic reactions attributed to compounds of similar chemical or biologic composition to study drug (e.g., rituximab or immunoglobulin G);
* Ongoing or active infection;
* Required the use of systemic antibiotics or antifungals for ongoing or recurrent infections. Topical use of antibiotics or antifungals is allowed;
* Other uncontrolled concurrent illness that would preclude study participation; or Psychiatric illness or social situation that would preclude study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Vonderheide, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States